CLINICAL TRIAL: NCT05085548
Title: A Phase I Trial of ProAgio, an Anti- αvβ3 Integrin Cytotoxin, for Previously Treated Advanced Pancreatic Cancer and Other Solid Tumor Malignancies
Brief Title: ProAgio in Previously Treated Advanced Pancreatic Cancer and Other Solid Tumor Malignancies
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ProDa BioTech, LLC (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 000194; 2R42CA217482-02 (NIH)
Record Dates: First submitted 2021-09-10; First posted 2021-10-20 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Advanced Pancreatic Cancer; Solid Tumor Malignancies

STUDY DESIGN:
Intervention Model Description: This study includes a dose escalation arm, followed by an expansion arm at the ideal dose for participants with non-neuroendocrine pancreatic cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation (Experimental): Participants will receive ProAgio in escalating doses.
  Interventions: Drug: ProAgio Dose Levels (DL) 1,2,3; Drug: ProAgio Dose Levels (DL) 4,5,6; Drug: ProAgio Dose Levels 4a,5a,6a
- Expansion Biopsy Arm (Experimental): Pre- and post-treatment tumor biopsy is optional for participants enrolled in the standard arm, but mandatory for participants enrolled in the biopsy arm.
  Interventions: Drug: ProAgio Dose Levels 4a,5a,6a
- Standard Arm (Experimental): Participants will receive ProAgio at the RP2D and may elect to receive concurrent gemcitabine beginning with the start of Cycle 2.
  Interventions: Drug: ProAgio Dose Levels (DL) 4,5,6; Drug: ProAgio Dose Levels 4a,5a,6a

INTERVENTIONS:
Drug: ProAgio Dose Levels (DL) 1,2,3 — ProAgio is administered to study participants by intravenous injections once every 14 days.
  Other Names: ACT50
  Arms: Dose Escalation
Drug: ProAgio Dose Levels (DL) 4,5,6 — ProAgio is administered to study participants by intravenous injections once every 7 days.
  Other Names: ACT50
  Arms: Dose Escalation; Standard Arm
Drug: ProAgio Dose Levels 4a,5a,6a — ProAgio is administered to study participants by intravenous injections once every 7 days with a drug holiday after every 5 administrations. Optional co-administration of gemcitabine (Gem) during dose expansion beginning with Cycle 2.
  Other Names: ACT50; Gemcitibine

SUMMARY:
The study is a first-in-human, Phase I study to assess the safety of ProAgio in participants with advanced solid tumor malignancies including pancreatic cancer.

DETAILED DESCRIPTION:
Pancreatic cancer is the third leading cause of death from cancer in the United States. The median overall survival for patients with metastatic disease who are receiving the most effective combination of chemotherapy regimens remains less than 1 year.

ProAgio has been evaluated in nonclinical pharmacology, safety pharmacology, pharmacokinetic (PK), and toxicity studies. It has demonstrated efficacy at treating pancreatic cancer and prolonging survival in mice.

ProAgio is being developed for intravenous (IV) administration. All participants will receive ProAgio until disease progression, unacceptable toxicity, or withdrawal from study. Subjects in the dose escalation cohorts who will be administered ProAgio at doses ranging from 3.2 to 36.8 mg/kg.

Following the dose escalation phase, an expansion cohort of patients with advanced nonendocrine pancreatic adenocarcinoma will be administered ProAgio at the maximum tolerated dose (MTD) from the dose escalation phase. Patients will also be offered optional co-administration of gemcitabine (Gem). The expansion cohort will contain two arms: A) Biopsy Arm (8 participants), and B) Standard Arm (8 participants). Tumor biopsies performed pre- and post- (on Cycle 2 Day 2-3) ProAgio treatment are optional for participants enrolled in the Standard Arm, but mandatory for participants enrolled in the Biopsy Arm.

ELIGIBILITY:
Inclusion Criteria:

For the Escalation Cohort:

* Histologic or cytologic diagnosis of a solid tumor malignancy for which no curative therapy exists.
* Individuals must have evaluable disease, either by clinical exam, biochemical markers (including but not limited to CA 19-9 serum tumor marker for pancreatobiliary cancer, or other appropriate tumor marker in other tumor types), and/or radiographic studies.
* Individuals must have received at least one prior systemic treatment for advanced disease.
* For the Expansion Cohort:
* Histologic or cytologic diagnosis of non-neuroendocrine pancreatic cancer. Individuals with mixed acinar-neuroendocrine histology are eligible.
* All Participants must have measurable disease, per RECIST 1.1.
* All individuals must have advanced or recurrent disease and have received at least one prior systemic treatment. Specifically:

  * Individuals with metastatic, locally advanced/unresectable, or borderline resectable pancreatic cancer at diagnosis, must have received at least one prior systemic treatment and still be considered ineligible for potentially curative resection.
  * Individuals who have undergone surgical resection and have tumor recurrence that is not amenable to local therapy, are eligible if:
* Tumor recurs within six months of the completion of adjuvant therapy, OR
* Further standard of care therapy is not a viable option due to prior resistance or intolerance, or a medical contraindication to both FOLFIRINOX (or NALIRIFOX) and gemcitabine-based chemotherapy
* Individuals in the Biopsy Arm of the expansion cohort must have disease amenable to safe biopsy and willingness to undergo the procedure.
* All individuals must be more than 14 days removed from most recent standard of care or experimental drug treatment for their tumor.
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of ProAgio in individuals <18 years of age, children are excluded from this study.
* ECOG performance status ≤ 2 (Karnofsky ≥>60%).
* Individuals must have adequate organ and marrow function as defined below:
* Aabsolute neutrophil count (ANC) ≥1,000/mcL
* hemoglobinHemoglobin (hgb) ≥9 g/ dL
* plateletsPlatelets ≥75,000/mcL
* Aspartate aminotransferase (AST)/ alanine transaminase (ALT) ( ≤ 2.5 x institutional upper limit of normal (ULN). AST and ALT (up to 5x ULN) is permitted for participants individuals with liver metastases)
* Total bilirubin ≤1.5 X institutional ULN
* Creatinine within normal institutional limits OR
* creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above institutional normal
* Serum albumin >2.5 mg/dL without intravenous supplementation
* Individuals must also have:
* Baseline QTcF interval of ≤ 470 ms
* Baseline resting heart rate > 45 beats per minute and <100 beats per minute
* Individuals of child-bearing potential (IOCBP) and individuals able to father a child men must agree to use an effective method of contraception as follows:
* IOCBP must agree to use an effective method of contraception (barrier, surgical sterilization, abstinence) prior to study entry, for the duration of study participation, and for at least 6 months after the last dose of study drug(s).
* Individuals able to father a child must agree to use an effective method of contraception (barrier, surgical sterilization, abstinence) for the duration of the study treatment and up to 6 months after the last dose of the study drug(s). We also will recommend individuals able to father a child with IOCBP partners to ask them to be on an effective birth control (hormonal, intrauterine device [(IUD)], surgical sterilization.
* Ability of individual to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Diagnosis of primary malignant CNS tumor.
* Individuals who are receiving any other investigational agents.
* Evidence of significant, uncontrolled concomitant diseases which could affect compliance with the protocol or interpretation of results, including but not limited to significant pulmonary disease other than that related to the primary cancer, uncontrolled diabetes mellitus, unstable angina, significant cardiovascular disease (such as New York Heart Association Class III or IV cardiac disease) and/or psychiatric illness/social situations within 12 weeks that would limit compliance with study requirements.
* Individuals with known diagnosis of a chronic neurologic disorders (such as multiple sclerosis, Huntington's disease, Parkinson's disease, or uncontrolled epilepsy) which causes motor disturbance, visual disturbance or seizure and could confound assessment of neurologic toxicity caused by the study drug.
* Pregnant or nursing individuals are excluded from this study because ProAgio is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with ProAgio, breastfeeding should be discontinued if the mother is treated with ProAgio.
* Individuals with leptomeningeal disease or with CNS metastases that are untreated, have required steroid treatment within the last 4 weeks, or anti-convulsant therapy in the last 14 days. For dose escalation cohort only: Individuals with any known CNS metastases are excluded. Those with symptoms suggestive of possible CNS metastases (such as new headaches) must undergo brain MRI as part of screening.
* Individuals who have undergone a recent minor surgical procedure (within <14 days) such as biliary stenting or major surgical procedure (within ≥ 28 days).
* Individuals who have undergone recent (within ≤ 14 days) external beam radiation therapy are excluded. Individuals who have undergone recent (within ≤ 28 days) treatment with radioactive therapeutics (such as Y90 or radio-immune conjugates) are ineligible.
* Individuals with uncontrolled bleeding episodes <28 days prior to enrollment are excluded.
* Individuals with active or uncontrolled infections are excluded.
* Individuals with HIV and detectable viral load are excluded. Patents on appropriate highly active anti-retroviral therapy with undetectable viral load are eligible.
* Individuals with a history of Hepatitis B or C are excluded unless there is documented evidence of effective treatment and/or cure with undetectable viral load.
* Individuals with recent (within < 28 days) thromboembolic disease including but not limited to acute coronary syndrome, stroke, or transient ischemic attack, recent deep vein thrombosis or pulmonary embolism.
* Individuals with thromboembolic disease including but not limited to acute coronary syndrome, stroke, or transient ischemic attack, recent deep vein thrombosis or pulmonary embolism who have continued symptoms, or who are not on stable doses of appropriate antiplatelet / anticoagulant regimens are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-10-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Determine Recommended Phase 2 Dose (RP2D) | 3 Years
  Following completion of the dose escalation cohort, all available data relating to the pharmacokinetics, pharmacodynamics, efficacy and safety of ProAgio will be reviewed by the study team including the Principle Investigator, clinical pharmacology collaborators and the sponsor. A single ideal dose will then be selected for further investigation in the dose escalation cohort. This ideal dose may or may not be the same as the MTD.

SECONDARY OUTCOMES:
Safety and Tolerability of ProAgio | 3 Years
  Toxicities will be tabulated and reported per dose level according to grade and type of toxicity experienced. This will take place during the dose escalation phase as well as during the expansion phase.
Evaluate the Maximum Plasma Concentration of ProAgio | 3 Years
  ProAgio concentrations will be measured by a validated ELISA assay modified from the assay used in non-clinical studies. This PK data will be used to mathematically describe the kinetic disposition of ProAgio in humans following the current dosing schedule.
Evaluate the area under the curve of ProAgio | 3 Years
  Statistical analysis of study data will calculate the area under the plasma concentration curve for each study subject that received ProAgio.
Evaluate the Serum half-life of ProAgio | 3 Years
  ProAgio Serum half-life will be determined using standard statistical calculations. .
Evaluate the volume of distribution of ProAgio | 3 Years
  If there are sufficient participant data available, a population PK analyses will be conducted to identify covariates that may be significantly associated with the inter-individual variability for a particular PK parameter (e.g. clearance of volume of distribution).The NCI CPP may also conduct dose-response and/or exposure-response analyses that will assess PK/PD relationships with relevant biomarkers, clinical response, and adverse event data.
Rate of study drug elimination in research participants | 3 Years
  58 study participants will have study drug concentration levels analyzed with regard to drug elimination. Results will be expressed in units of inverse time, i.e. 1/hr or 1/day.
Objective Response Rate (ORR) | 3 Years
  Make a preliminary assessment of anti-tumor activity by measuring objective response rate (ORR),
Disease control rate (DCR). | At 18 Weeks
  Make a preliminary assessment of anti-tumor activity by measuring disease control rate at 18 weeks (DCR).
Assess serum tumor marker CA19-9 or appropriate tumor specific marker. | Day 1 of each treatment cycle and 30 days after the last dose of study therapy.
  Make a preliminary assessment of anti-tumor activity by measuring change in relevant serum tumor marker CA19-9 appropriate tumor specific marker.

OTHER OUTCOMES:
Assess whether a host antibody response against ProAgio develops with repeated administration | 2 Years
  Change in ADA titer, as measured between baseline and EOT
Assess biologic effect of ProAgio on apoptosis of tumor cells in tumor tissue | 2 Years
  Pre- to on-therapy tumor biopsy specimen assessment of changes in apoptosis of tumor cells
Assess biologic effect of ProAgio on integrin αvβ3 expression in tumor tissue | 2 Years
  Pre- to on-therapy tumor biopsy specimen assessment of changes in integrin αvβ3 expression (% of cells expressing both integrins)
Assess biologic effect of ProAgio on tumor collagen density and architecture | 2 Years
  Pre- to on-therapy tumor biopsy specimen assessment of changes in tumor collagen density and architecture (Sirius Red stain)
Assess biologic effect of ProAgio on tumor vasculature | 2 Years
  Pre- to on-therapy tumor biopsy specimen assessment of changes in tumor vasculature (% of CD31 positive cells)
Assess biologic effect of ProAgio on CAF and CASCs populations | 2 Years
  Pre- to on-therapy tumor biopsy specimen assessment of changes on CAF and CASCs populations (% of α-SMA positive cells)
Assess biologic effect of ProAgio on changes on Localization / populations of tumor cells | 2 Years
  Pre- to on-therapy tumor biopsy specimen assessment of changes on Localization / populations of tumor cells as measured by Digital spatial profiling (DSP)
Identify surrogate circulating biomarkers of ProAgio bioactivity in serum PKM2 concentrations | 2 Years
  Pre- to on-therapy change in serum PKM2 concentration
Identify surrogate circulating biomarkers of ProAgio bioactivity in CECs quantities | 2 Years
  Pre- to on-therapy change in CECs quantities
Identify surrogate circulating biomarkers of ProAgio bioactivity on circulating fibroblasts quantities | 2 Years
  Pre- to on-therapy change on circulating fibroblasts quantities
Identify surrogate circulating biomarkers of ProAgio bioactivity in Circulating αvβ3 expressing cells | 2 Years
  Pre- to on-therapy change in Circulating αvβ3 expressing cells (all cells and CTCs)
Assess the safety of co-administering ProAgio with gemcitabine (Gem) | 2 Years
  For cycles where participants receive both ProAgio and Gem, tabulated list of:
  * Grade ≥ 3 and higher adverse events (AEs)
  * All AEs attributable to research
  * Whether or not stopping rules for optional addition of Gem are met
Evaluate maximum plasma concentration (Cmax) of ProAgio when given in combination with Gem | 2 Years
  For cycles where participants receive both ProAgio and Gem determine maximum plasma concentration (Cmax)
Evaluate serum half-life of ProAgio when given in combination with Gem | 2 Years
  For cycles where participants receive both ProAgio and Gem estimate serum half-life

CONTACTS AND LOCATIONS:
Overall Officials: Anish Thomas, MBBS, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No